CLINICAL TRIAL: NCT01506427
Title: A Phase I/II, Open Label, Nonrandomized, Multi-Center Study of [F-18]HX4 Positron Emission Tomography (PET) in Head and Neck Cancer Patients
Brief Title: A Study of [F-18]HX4 (PET Imaging)Evaluated in Head and Neck Cancer Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Siemens Molecular Imaging (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HX4-201
Record Dates: First submitted 2011-12-28; First posted 2012-01-10 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Head and Neck Cancer
Keywords: Newly Diagnosed; Head and Neck Cancer; PET Imaging
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [F-18] HX4 (Experimental)
  Interventions: Radiation: [F-18] HX4

INTERVENTIONS:
Radiation: [F-18] HX4 — A single dose of 10 mCi, injected intravenously.

SUMMARY:
The purpose of this trial is to determine what will be the optimal imaging protocol for Head and Neck Cancer patients after [F-18] HX4 injection. This study will provide guidance for future studies involving [F-18]HX4 in cancer patients.

DETAILED DESCRIPTION:
Each consented patient will have a single administration of [F-18]HX4 and will immediately undergo one list mode PET/CT imaging session lasting 60 minutes followed by three additional list mode PET/CT acquisitions from 90 to 110 minutes, 150 to 170 minutes and 220 to 250 minutes after administration. The start times of the last three image acquisitions are permitted to be within ± 5 minutes. Venous blood samples will be collected throughout the initial scan sequence and at the time of each subsequent acquisition for calibration and metabolite-correction of the image-derived input function. On the day of administration (Visit 2) blood for clinical safety evaluations will be drawn pre- and post-dosing after all imaging is complete.

The pre-surgery [F-18]FDG PET/CT clinical scan performed prior to the [F-18]HX4 procedure, and the surgery at Visit 3 are standard of care for the consented patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is >18 years and male or female of any race / ethnicity.
* Patient or patient's legally acceptable representative provides written inform consent Patient is willing and able to comply with protocol procedures.
* Patient has newly diagnosed histologically confirmed squamous cell carcinoma of the head and/or neck whose primary origin is from the oral cavity, oropharynx, hypopharynx, larynx or nasopharynx.
* Patient is scheduled to have or already has had a clinical [F-18]FDG PET/CT scan prior (recommended to be within 14 days prior) to the [F-18]HX4 PET/CT scan.
* Patient has a primary tumor ≥ 2.0 cm in longest axis measured by CT or MR; or lymph node ≥ 2.0 cm in shortest axis measured by CT or MR if primary tumor < 2 cm on CT or MR; CT may be part of required [F-18]FDG PET/CT scan or a separate pre-surgery CT scan.
* Patient is scheduled to undergo complete tumor resection within 7 days for his/her cancer care after the [F-18]HX4 PET/CT scan is performed.
* Patient has not had nor will have neoadjuvant treatment, including radiation and chemotherapy, prior to patient's planned tumor resection.

Exclusion Criteria:

* Female patient is pregnant or nursing.
* Patient is not capable of remaining still for duration of imaging procedure (~ 4 hours).
* Patient has undergone an investigative, radioactive research procedure within 7 days prior to study participation, or is scheduled to undergo such a procedure during the study participation period.
* Patient has chronic renal function failure or is on renal dialysis
* Patient has any other condition or personal circumstance that, in the judgment of the investigator, might interfere with the collection of complete data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2013-04 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Serial measures of T/B Ratios and other imaging parameters | Approximately 1 month after patient imaging; comprehensive analysis will be concluded within 1 month after Last Patient Out
  Serial measures of T/B ratios and other imaging parameters derived from the course imaging data of head and neck cancer pateitns in order to determine time of optimal imaging.

SECONDARY OUTCOMES:
Correlations between T/B ratios of [F-18]HX4 uptake from pre-surgery PET imaging and immunohistochemistry measurements | Estimated analysis to occur 1 month after patient surgery
  Correlations between T/B ratios of [F-18]HX4 uptake from pre-surgery PET imaging and immunohistochemistry measurements obtained from surgical tumor samples
Kinetic Modeling Analysis | Estimated to be 2 weeks after the Imaging Date (Visit 2)
  Kinetic parameters obtained from modeling time course of PET imaging data following [F-18]HX4 administration
Safety Assessments | On average of 3 weeks (from Time of Signing Consent to 24 hours after the Imaging Date)
  Safety measurements including incidence of adverse events, and pre- and post-drug clinical laboratory measurements, vital signs and electrocardiograms

CONTACTS AND LOCATIONS:
Overall Officials: John Buatti, MD, Principal Investigator — University of Iowa Medical Center; Edward Aten, MD, Study Director — President, Certus International
Locations (1):
- University of Iowa Medical Center, Iowa City, Iowa, United States